CLINICAL TRIAL: NCT02094885
Title: A Prospective, Randomized, Controlled Phase IV Study to Compare Bioseal Versus Manual Compression as an Adjunct to Hemostasis in the Patients Undergoing Elective Vascular Surgery
Brief Title: The Bioseal Vascular Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: Guangzhou Bioseal Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS-13-003
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Bleeding; Vascular Bleeding; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioseal Fibrin Sealant (Experimental): A porcine-derived fibrin sealant consisting of thrombin and fibrinogen
  Interventions: Biological: Bioseal Fibrin Sealant
- Manual compression (Other): Manual compresssion (MC) include any active or inactive adjunctive treatment to hemostasis methods currently used based on each surgeons surgical practice except for the use of other fibrin sealants.
  Interventions: Other: Manual Compression

INTERVENTIONS:
Biological: Bioseal Fibrin Sealant
  Arms: Bioseal Fibrin Sealant
Other: Manual Compression
  Arms: Manual compression

SUMMARY:
To evaluate the clinical utility of Bioseal as an adjunct to control bleeding during elective vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18 and 75 years of age;
2. Undergoing elective vascular surgical procedures and with the presence of an appropriate Target Bleeding Site (TBS) requiring an adjunct to achieve hemostasis as identified intra-operatively by the surgeon ;
3. Able and willing to comply with procedures required by protocol;
4. Signed and dated written informed consent prior to any study related procedures.

Exclusion Criteria:

1. Subjects with any intra-operative findings that may preclude conducting of the study procedures;
2. Intended use of Fibrin Sealants (including autologous Fibrin Sealants) other than Bioseal on the TBS;
3. Subjects with known intolerance to blood products or to one of the components of the study product or unwilling to receive blood products;
4. Subjects with known allergies to or previously used porcine derived products;
5. Female subjects who are known breastfeeding or pregnant or intend to become pregnant during the clinical study period.
6. The subject, in the opinion of the investigator, would not be suitable for participation in the study.
7. Subjects who participated in another trial within 30 days prior to the planned start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (9):
- China (9):
  - Clinical Investigation Site #21, Guangzhou, Guangdong
  - Clinical Investigation Site #32, Nanjing, Jiangsu
  - Clinical Investigation Site #31, Nanjing, Jiangsu
  - Clinical Investigation Site #30, Jinan, Shandong
  - Clinical Investigation Site #22, Chengdu, Sichuan
  - Clinical Investigation Site #26, Beijing
  - Clinical Investigation Site #28, Beijing
  - Clinical Investigation Site #25, Shanghai
  - Clinical Investigation Site #23, Shanghai

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Compression: Manual compression (MC) include any active or inactive adjunctive treatment to hemostasis methods currently used based on each surgeons surgical practice except for the use of other fibrin sealants.
Period: Overall Study
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Started | 125 | 127
Completed | 123 | 122
Not Completed | 2 | 5
Not completed — Death | 1 | 5
Not completed — Withdrawn due to age | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bioseal Fibrin Sealant | Manual Compression | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.0) | 56.8 (12.2) | 56.9 (12.6)
Age, Customized [Number; unit: Participants]
  <=60 years | 63 | 64 | 127
  >60,<=75 years | 60 | 63 | 123
  >75 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 90 | 94 | 184
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (3.4) | 23.8 (3.2) | 23.9 (3.3)
BMI Group [Number; unit: participants] — BMI Categories:
  Underweight: <18.5 lb/inch^2; Normal: 18.5<=BMI<25; Overweight: 25<=BMI<30 Obese: 30<=BMI<40 Morbidly obese: BMI>=40
  participants
    Underweight | 6 | 6 | 12
    Normal | 75 | 79 | 154
    Overweight | 41 | 39 | 80
    Obese | 3 | 3 | 6
Height [Mean (Standard Deviation); unit: cm] | 167.2 (7.0) | 166.6 (7.8) | 166.9 (7.4)
Height [Median (Full Range); unit: cm] | 168.0 [152.0 to 190.0] | 167.0 [145.0 to 186.0] | 168.0 [145.0 to 190.0]
Weight [Mean (Standard Deviation); unit: kg] | 67.1 (11.6) | 66.3 (11.2) | 66.7 (11.4)
Weight [Median (Full Range); unit: kg] | 67.0 [40.0 to 95.0] | 66.0 [45.0 to 100.0] | 66.0 [40.0 to 100.0]
Smoking Status [Number; unit: participants]
  Current Smoker | 39 | 31 | 70
  Former Smoker | 15 | 17 | 32
  Never Smoked | 71 | 79 | 150

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 10 Minutes Following the Completion of Treatment Application.
Description: Percentage of participants with Hemostasis at the TBS at 10 minutes following the completion of treatment application. Hempstasis is defined as absence of bleeding.
Time Frame: Intra-operative, 10 minutes following randomization
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Number analyzed (Participants) | 125 | 127
percentage of patients | 96 [90.9 to 98.7] | 88.2 [81.3 to 93.2]

2. Secondary Outcome: Hemostasis at the Target Bleeding Site (TBS) at 3 and 6 Minutes Following the Completion of Treatment Application
Description: Percentage of participants with Hemostasis at the TBS at 3 and 6 minutes following the completion of treatment application. Hempstasis is defined as absence of bleeding.
Time Frame: Intra-operative, 3 and 6 minutes following randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Number analyzed (Participants) | 125 | 127
percentage of participants
  Hemostasis at 3 Minutes | 84 [76.4 to 89.9] | 43.3 [34.5 to 52.4]
  Hemostasis at 6 Minutes | 96.0 [90.9 to 98.7] | 74.0 [65.5 to 81.4]

3. Secondary Outcome: Number of Participants Requiring Alternative Treatment Due to Treatment Failure*
Description: Alternative treatments include the use of additional hemostatic methods, including collagen, manual compression, oxidized regenerated cellulose and suture. Manual compression (MC) may be applied after the initial 10 minute observation period as an alternative treatment due to treatment failure in either group. For participants with a treatment failure in MC group, the addition treatment of MC is applied after the initial 10 minute observation period.
Time Frame: Intra-operative, 10 minutes following randomization
Measure: Number; unit: participants
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Number analyzed (Participants) | 125 | 127
participants
  Total number requiring alternative treatment | 5 | 15
  Treated with Collagen | 0 | 2
  Treated with Manual Compression After 10 Minutes* | 1 | 1
  Treated with Oxidized Regenerated Cellulose | 2 | 8
  Treated with Suture | 2 | 4

4. Secondary Outcome: Percentage of Participants With Potential Bleeding-related Adverse Events
Description: Percentage of participants with potential bleeding-related adverse events by study group
Time Frame: 30-days follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Number analyzed (Participants) | 125 | 127
percentage of participants | 2.4 [0.5 to 6.9] | 2.4 [0.5 to 6.7]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of randomization during the procedure until completion of the 30 day follow-up visit.
Arm/Group | Bioseal Fibrin Sealant | Manual Compression
Serious Adverse Events (participants affected / at risk) | 13/125 | 11/127
Other Adverse Events (participants affected / at risk) | 15/125 | 13/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bioseal Fibrin Sealant (N=125) | Manual Compression (N=127)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial Rupture (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ Failure (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Livery Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Post-procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acinetobacter Test Positive (Investigations) | 1 (1) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic Dissection Rupture (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bioseal Fibrin Sealant (N=125) | Manual Compression (N=127)
Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less